CLINICAL TRIAL: NCT06290258
Title: Fecal Microbiota Transplantation for Gastrointestinal, Autistic, Emotion, and Behavior Symptoms of Patients With Autism Spectrum Disorder and Gastrointestinal Problems: a Preliminary Study.
Brief Title: Fecal Microbiota Transplantation for Patients With Autism Spectrum Disorder.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202202143A0
Record Dates: First submitted 2024-01-31; First posted 2024-03-04 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder; Gastrointestinal Diseases; Healthy
Keywords: Fecal Microbiota Transplantation; Autism Spectrum Disorder; gastrointestinal problems; cytokines; cognitive function
MeSH Terms: conditions — Autism Spectrum Disorder; Gastrointestinal Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal microbiota transplantation (Experimental): Children with autism spectrum disorder will receive fecal microbiota transplantation after evaluation. After the first intervention, the second transplantation will be arranged 6 months later.
  Interventions: Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Fecal microbiota transplantation has been applied to patients with autism spectrum disorder in recent years. Fecal microbiota of healthy donors can be transplanted to patients through colonoscopy. Before donation, donors were comprehensively screened to rule out gastrointestinal symptoms and infections. Patients will receive colon preparation before transplantation. After the intervention, patients will have to stay in bed and be monitored for 24 hours to assure safety.

SUMMARY:
This study aims to evaluate the efficacy of fecal microbiota transplantation on the gastrointestinal symptoms, autistic symptoms and emotional behavior symptoms of patients with autism spectrum disorder, and investigate the relations between the brain-gut axis, cytokines and autism spectrum disorder. Fecal microbiota transplantation have the potentials to improve intestinal microbiota composition, regulate immunity, and then improve gastrointestinal symptoms, autistic symptoms, emotional behavior symptoms and sleep of children with autism spectrum disorder. Early intervention at school-age may even benefit development, improve cognition and prognosis.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is an early neuropsychiatric developmental disorder. About 7-90% of patients with ASD have gastrointestinal problems which can relate to abnormal intestinal microbiota. The brain-gut axis can play a key role in the development of brain, and the interaction between microbiota and central nerve system can relate to the pathophysiology of ASD. Fecal Microbiota Transplantation (FMT) has just been used in the treatment of ASD in recent years. It has the potential to improve gastrointestinal, autistic, emotion and behavior symptoms of patients with ASD. Studies of its efficacy are still scarce, and no study has been conducted in Taiwan.

The purpose of this study is to treat patients with ASD by the fecal microbiota transplantation and evaluate its efficacy in gastrointestinal, autistic, emotion and behavior symptoms. It aims to prove the correlations between the brain-gut axis, intestinal microbiota, cytokines and ASD. FMT may improve and change the composition and diversity of intestinal microbiota of patients with ASD and modulate their immune reactions and subsequently improve gastrointestinal, autistic, emotion and behavior symptoms, as well as sleep. Early intervention by FMT in children with ASD may improve their cognition and hence result in better prognosis.

Study design: The investigators will recruit 45 patients with ASD and gastrointestinal problems, aged 6-30 years, who are willing to receive FMT and 1-year regular follow-up. The investigators will collect demographic data, blood and stool samples before and after the intervention, and analyze changes of intestinal microbiota and cytokines. The investigators will use subjective questionnaires to evaluate gastrointestinal, autistic, emotion and behavior symptoms, and objective measurements including actigraphy, intelligence and attention tests to evaluate changes in sleep and cognitive functions. The investigators will analyze the correlations between collected variables and compare the ASD group with the healthy control group at baseline to evaluate group differences. The investigators will evaluate the differences of the intervention group before and after FMT, and also compare the intervention group with the waiting list group, to evaluate the efficacy of FMT. Variables will be presented by mean and percentage. The investigators will use independent sample t-test or Chi-squared test for group comparison. The efficacy of FMT will be analyzed by dependent sample t-test or Wilcoxon signed-rank test, and the investigators will use Pearson correlation coefficient to analyze the correlations between variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by a child psychiatrist in line with DSM-5 Autism Spectrum Disorder
* Combined with gastrointestinal problems, any Gastrointestinal Symptoms Rating Scale score≧3.
* Age is between 7-30.
* Participants who are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Cases where clinical assessment cannot cooperate with fecal microbiota transplantation and examination.
* Cases requiring antibiotics within 3 months before or after acceptance because of their physiological condition.
* Cases requiring long-term use of proton pump inhibitors due to their physiological conditions.
* Severe physical diseases, such as acute gastrointestinal diseases, severe malnutrition or underweight, immunodeficiency diseases, severe allergies or autoimmune diseases, brain injuries or severe organic brain diseases, will affect the evaluation of treatment results.
* Severe mental illness, such as schizophrenia, bipolar disorder, etc.
* Those who used probiotics one month before the case may affect the intestinal flora.
* Pregnancy.
* Cases that cannot understand the content of this research.
* Participants who are unwilling to participate in the study or refuse to sign the informed consent.
* Participants who are not suitable to include in this study, evaluate by PI or Co-PI.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes of gastrointestinal symptoms of patients with ASD after FMT | baseline and the 1-year follow-up
  the Gastrointestinal Symptom Rating Scale, score 15-105, higher scores mean more severe symptom
Changes of autistic symptoms of patients with ASD after FMT | baseline and the 1-year follow-up
  the Social Responsiveness Scale, score 0-195, higher scores mean more severe symptom

SECONDARY OUTCOMES:
Changes of the diversity of intestinal microbiota of patients with ASD after FMT | baseline and the 1 year follow-up
  microbial DNA was extracted from feces by Reagent Kit v3, and the diversity indices were calculated by using the vegan package in R version 3.2.3. higher indices suggest higher microbial diversity
Changes of cytokine levels of patients with ASD after FMT | baseline and the 1 year follow-up
  cytokine levels
Changes of repetitive behavior symptoms of patients with ASD after FMT | baseline and the 1 year follow-up
  the Repetitive Behavior Scale-Revised data, higher score suggest more repetitive behavior
Changes of autistic behavior symptoms of patients with ASD after FMT | baseline and the 1 year follow-up
  the Aberrant Behavior Checklist data, higher score suggest more autistic behavior
Changes of emotion and behavior symptoms of patients with ASD after FMT | baseline and the 1 year follow-up
  the Child Behavior Checklist Adaptive Behavior Assessment System® - Second Edition data, higher score suggest more emotion and behavior symptoms
Changes of inattention and hyperactivity of patients with ASD after FMT | baseline and the 1 year follow-up
  the Swanson, Nolan and Pelham IV Scale data, higher score suggest worse attention and more hyperactivity
Changes of quality of life of patients with ASD after FMT | baseline and the 1 year follow-up
  the 36-Item Short Form Health Survey data, higher score suggest better quality of life

OTHER OUTCOMES:
Changes of objective sleep of patients with ASD after FMT by actigraphy recording | baseline and the 1 year follow-up
  Participants wear actigraphy for 7-10 days to record their activities and light exposure, which can be calculated to represent their sleep patterns. Sleep parameters including (total sleep time: minutes, sleep efficiency: percentage, total time in bed: minutes, sleep onset latency: minutes, wakefulness after sleep onset: minutes, the sum of wake duration overnight: minutes, total number of awakenings: times, sleep onset time and wake time: hours and minutes) will be obtained and analyzed.
Changes of subjective sleep of patients with ASD after FMT | baseline and the 1 year follow-up
  the Children's Sleep Habits Questionnaire data, higher score suggest poorer sleep
Changes of intelligence of patients with ASD after FMT | baseline and the 1 year follow-up
  the Wechsler Intelligence Scale data, higher score suggest better intelligence
Changes of attention and impulse control of patients with ASD after FMT | baseline and the 1 year follow-up
  the Conners' Continuous Performance Test data, higher score suggest worse attention and impulse control

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chih Chin, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Wei-Chih Chin, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams JB, Johansen LJ, Powell LD, Quig D, Rubin RA. Gastrointestinal flora and gastrointestinal status in children with autism--comparisons to typical children and correlation with autism severity. BMC Gastroenterol. 2011 Mar 16;11:22. doi: 10.1186/1471-230X-11-22. PMID 21410934
- [Background] Alharthi A, Alhazmi S, Alburae N, Bahieldin A. The Human Gut Microbiome as a Potential Factor in Autism Spectrum Disorder. Int J Mol Sci. 2022 Jan 25;23(3):1363. doi: 10.3390/ijms23031363. PMID 35163286
- [Background] Ashwood P, Krakowiak P, Hertz-Picciotto I, Hansen R, Pessah I, Van de Water J. Elevated plasma cytokines in autism spectrum disorders provide evidence of immune dysfunction and are associated with impaired behavioral outcome. Brain Behav Immun. 2011 Jan;25(1):40-5. doi: 10.1016/j.bbi.2010.08.003. Epub 2010 Aug 10. PMID 20705131
- [Background] Baldi S, Mundula T, Nannini G, Amedei A. Microbiota shaping - the effects of probiotics, prebiotics, and fecal microbiota transplant on cognitive functions: A systematic review. World J Gastroenterol. 2021 Oct 21;27(39):6715-6732. doi: 10.3748/wjg.v27.i39.6715. PMID 34754163
- [Background] Baxter M, Colville A. Adverse events in faecal microbiota transplant: a review of the literature. J Hosp Infect. 2016 Feb;92(2):117-27. doi: 10.1016/j.jhin.2015.10.024. Epub 2015 Dec 15. PMID 26803556
- [Background] Borre YE, O'Keeffe GW, Clarke G, Stanton C, Dinan TG, Cryan JF. Microbiota and neurodevelopmental windows: implications for brain disorders. Trends Mol Med. 2014 Sep;20(9):509-18. doi: 10.1016/j.molmed.2014.05.002. Epub 2014 Jun 20. PMID 24956966
- [Background] Croonenberghs J, Bosmans E, Deboutte D, Kenis G, Maes M. Activation of the inflammatory response system in autism. Neuropsychobiology. 2002;45(1):1-6. doi: 10.1159/000048665. PMID 11803234
- [Background] Hsiao EY, McBride SW, Hsien S, Sharon G, Hyde ER, McCue T, Codelli JA, Chow J, Reisman SE, Petrosino JF, Patterson PH, Mazmanian SK. Microbiota modulate behavioral and physiological abnormalities associated with neurodevelopmental disorders. Cell. 2013 Dec 19;155(7):1451-63. doi: 10.1016/j.cell.2013.11.024. Epub 2013 Dec 5. PMID 24315484
- [Background] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648
- [Background] Kang DW, Adams JB, Coleman DM, Pollard EL, Maldonado J, McDonough-Means S, Caporaso JG, Krajmalnik-Brown R. Long-term benefit of Microbiota Transfer Therapy on autism symptoms and gut microbiota. Sci Rep. 2019 Apr 9;9(1):5821. doi: 10.1038/s41598-019-42183-0. PMID 30967657
- [Background] Li N, Chen H, Cheng Y, Xu F, Ruan G, Ying S, Tang W, Chen L, Chen M, Lv L, Ping Y, Chen D, Wei Y. Fecal Microbiota Transplantation Relieves Gastrointestinal and Autism Symptoms by Improving the Gut Microbiota in an Open-Label Study. Front Cell Infect Microbiol. 2021 Oct 19;11:759435. doi: 10.3389/fcimb.2021.759435. eCollection 2021. PMID 34737978
- [Background] McElhanon BO, McCracken C, Karpen S, Sharp WG. Gastrointestinal symptoms in autism spectrum disorder: a meta-analysis. Pediatrics. 2014 May;133(5):872-83. doi: 10.1542/peds.2013-3995. PMID 24777214
- [Background] Molloy CA, Morrow AL, Meinzen-Derr J, Schleifer K, Dienger K, Manning-Courtney P, Altaye M, Wills-Karp M. Elevated cytokine levels in children with autism spectrum disorder. J Neuroimmunol. 2006 Mar;172(1-2):198-205. doi: 10.1016/j.jneuroim.2005.11.007. Epub 2005 Dec 19. PMID 16360218
- [Background] Samsam M, Ahangari R, Naser SA. Pathophysiology of autism spectrum disorders: revisiting gastrointestinal involvement and immune imbalance. World J Gastroenterol. 2014 Aug 7;20(29):9942-51. doi: 10.3748/wjg.v20.i29.9942. PMID 25110424
- [Background] Souders MC, Mason TB, Valladares O, Bucan M, Levy SE, Mandell DS, Weaver TE, Pinto-Martin J. Sleep behaviors and sleep quality in children with autism spectrum disorders. Sleep. 2009 Dec;32(12):1566-78. doi: 10.1093/sleep/32.12.1566. PMID 20041592
- [Background] Strati F, Cavalieri D, Albanese D, De Felice C, Donati C, Hayek J, Jousson O, Leoncini S, Renzi D, Calabro A, De Filippo C. New evidences on the altered gut microbiota in autism spectrum disorders. Microbiome. 2017 Feb 22;5(1):24. doi: 10.1186/s40168-017-0242-1. PMID 28222761
- [Background] Tan Q, Orsso CE, Deehan EC, Kung JY, Tun HM, Wine E, Madsen KL, Zwaigenbaum L, Haqq AM. Probiotics, prebiotics, synbiotics, and fecal microbiota transplantation in the treatment of behavioral symptoms of autism spectrum disorder: A systematic review. Autism Res. 2021 Sep;14(9):1820-1836. doi: 10.1002/aur.2560. Epub 2021 Jun 26. PMID 34173726
- [Background] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553
- [Background] Xu M, Xu X, Li J, Li F. Association Between Gut Microbiota and Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. Front Psychiatry. 2019 Jul 17;10:473. doi: 10.3389/fpsyt.2019.00473. eCollection 2019. PMID 31404299